CLINICAL TRIAL: NCT02167035
Title: Pilot Study Comparison of Combigan Two Times Daily (BID) vs Simbrinza Three Times Daily (TID) in Subjects Currently Treated With Latanoprost For Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Comparison of Combigan Two Times Daily (BID) Versus Simbrinza Three Times Daily (TID)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cornerstone Health Care, PA (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Michael Tepedino MD, Director of Clinical Research, Cornerstone Health Care, PA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEP001
Record Dates: First submitted 2014-06-12; First posted 2014-06-18 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combigan Two Times Daily (BID) (Active Comparator): Combigan 0.2%/0.5% one drop Two Times Daily (BID)
  Interventions: Drug: Combigan Two Times Daily (BID)
- Simbrinza Three Times Daily (TID) (Active Comparator): Simbrinza 1/0.2% one drop Three Times Daily (TID)
  Interventions: Drug: Simbrinza Three Times Daily (TID)

INTERVENTIONS:
Drug: Combigan Two Times Daily (BID)
  Arms: Combigan Two Times Daily (BID)
Drug: Simbrinza Three Times Daily (TID)
  Arms: Simbrinza Three Times Daily (TID)

SUMMARY:
To compare Combigan Two Times Daily (BID) vs Simbrinza Three Times Daily (TID) in subjects currently being treated with Latanoprost for Open-Angle Glaucoma or Ocular Hypertension. Both of these drugs are currently FDA approved as combination therapy for patients with Open-Angle Glaucoma or Ocular Hypertension. The purpose of this clinical trial would be to assess which treatment, if either, is superior in lowering intraocular pressure (IOP). A secondary objective is to assess the tolerability of each drug.

ELIGIBILITY:
Inclusion Criteria:

* Open-angle glaucoma or ocular Hypertension
* Currently treated with Latanoprost for min of 6 weeks
* Male or Female 18 yrs and older
* Best Corrected Visual Acuity 20/100 or better in both eyes
* Pachymetry >470 and < 640
* Women of childbearing potential must have a negative urine pregnancy test at the screening/baseline visit
* Patient willing and capable of providing informed consent

Exclusion Criteria:

* C/D > 0.8
* Visual field loss, which in the opinion of the investigator is functionally significant
* Current use of ocular steroids
* Concurrent significant active ocular disease History (within 3 months prior to Screening) of ocular laser, intraocular, filtering or refractive surgery or planned ocular surgery of any kind during study participation
* Change within prior 30 days or anticipated change in any systemic medication that is known to affect IOP
* Uncontrolled systemic disease
* Significant ocular hyperemia at baseline
* Prior glaucoma procedure within 3 months
* Females who are pregnant, nursing, or planning a pregnancy or who are of childbearing potential and not using a reliable method of contraception
* Known allergy or sensitivity to any study medication
* Asthma or any other known medical condition that the investigator feels would put patient at increased risk from any of the study medications
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Tepedino, MD, Principal Investigator — Cornerstone Health Care
Locations (1):
- Cornerstone Health Care, High Point, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Combigan Two Times Daily (BID): Combigan 0.2%/0.5% one drop Two Times Daily (BID)
  Combigan Two Times Daily (BID)
- Simbrinza Three Times Daily (TID): Simbrinza 1/0.2% one drop Three Times Daily (TID)
  Simbrinza Three Times Daily (TID)
Period: Overall Study
Arm/Group | Combigan Two Times Daily (BID) | Simbrinza Three Times Daily (TID)
Started | 21 | 22
Completed | 16 | 16
Not Completed | 5 | 6
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Randomized to incorrect Study Medication | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was conducted on the Safety Population (N=43) for Subject Demographics.
Groups:
- Combigan Twice Daily (BID): Combigan 0.2%/0.5% one drop Twice Daily (BID)
  Combigan Twice Daily (BID)
- Total: Total of all reporting groups
Arm/Group | Combigan Twice Daily (BID) | Simbrinza Three Times Daily (TID) | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (11.43) | 67.7 (8.43) | 67.8 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: The Intraocular Pressure will be assessed on study subjects. IOP (Intraocular Pressure) will be measured using a Goldmann applanation tonometer. Both eyes will be tested, with the right eye preceding the left eye. The operator will initially set the dial at 10 mmHg, then look through the slit lamp and adjust the dial to take the reading, and then record the results. The procedure will be repeated on the same eye twice consecutively. If the measurements are within 2mmHg or less of each other, the mean of the 2 reading will be reported as the IOP at that time point. If the 2 reading are more than 2mmHg apart from each other, a third (consecutive) reading will be taken and the median (middle) IOP will be reported as the IOP at that time point. Preferable, the same operator will measure IOP and the same tonometer will be used at each visit.
Time Frame: Day 0 (08:00, 10:00 16:00), Day 30 (08:00, 10:00, 16:00), Day 90 (08:00, 10:00,16:00)
Population: Primary endpoint analysis was conducted on the modified intent-to-treat (mITT) population, which consisted of all enrolled subjects randomized to masked study medication and who attended Visits 1,2,and 3 (minimally).
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Combigan BID: Combigan 0.2%/0.5% one drop Twice Daily (BID)
  Combigan Twice Daily (BID)
- Simbrinza TID: Simbrinza 1/0.2% one drop Three Times Daily (TID)
  Simbrinza Three Times Daily (TID)
Arm/Group | Combigan BID | Simbrinza TID
Number analyzed (Participants) | 17 | 19
mmHg
  Baseline 8am IOP | 19.7 (5.33) | 18.1 (3.31)
  Baseline 10am IOP | 19.1 (4.42) | 18.8 (4.26)
  Baseline 4pm IOP | 17.6 (4.24) | 17.6 (3.83)
  Baseline Diurnal IOP | 18.8 (4.42) | 18.1 (3.53)
  Visit 3 8am IOP | 17.6 (4.47) | 17.4 (2.26)
  Visit 3 10am IOP | 17.6 (3.08) | 16.2 (2.52)
  Visit 3 4pm IOP | 17.1 (3.36) | 17.6 (4.04)
  Visit 3 Diurnal IOP | 17.4 (3.12) | 17.0 (2.51)
  Visit 4 8am IOP | 18.7 (4.19) | 18.4 (3.44)
  Visit 4 10am IOP | 17.7 (3.33) | 18.1 (3.96)
  Visit 4 4pm IOP | 18.1 (3.22) | 17.6 (3.43)
  Visit 4 Diurnal IOP | 18.1 (2.66) | 18.0 (3.32)

2. Secondary Outcome: Ocular Symptom and Tolerability Questionaire
Description: The secondary endpoint of this study was to determine the tolerability of each treatment group by utilizing ocular symptom questionnaires administered at each study visit. These questionnaires assessed Oral effects (bad taste, dry mouth) and Ocular comfort effects (itching, burning, stinging, burning on instillation, blurred vision). The scale proved was none=0, mild=1, moderate=2, severe=3.
Time Frame: Baseline (Day 0), Visit 2 (Day 7), Visit 3 (Day 30), Visit 4 (Day 90)
Population: Secondary endpoint analysis was conducted on the modified intent-to-treat (mITT) population, which consisted of all enrolled subjects randomized to masked study medication and who attended Visits 1,2,and 3 (minimally).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Combigan BID: Combigan 0.2%/0.5% one drop BID
  Combigan BID
- Simbrinza TID: Simbrinza 1/0.2% one drop TID
  Simbrinza TID
Arm/Group | Combigan BID | Simbrinza TID
Number analyzed (Participants) | 17 | 19
units on a scale
  Baseline - Burning/Stinging Upon Instillation | 0.1 (0.33) | 0.1 (0.32)
  Baseline - non-instillation Burning/stinging | 0.1 (0.24) | 0.1 (0.32)
  Baseline - Dry/Gritty Eye | 0.3 (0.47) | 0.4 (0.60)
  Baseline - Foreign Body Sensation | 0.1 (0.24) | 0.1 (0.23)
  Baseline - Eye Redness | 0.1 (0.33) | 0.2 (0.63)
  Baseline - Blurred Vision | 0.1 (0.33) | 0.3 (0.56)
  Baseline - Dry Mouth | 0.2 (0.53) | 0.0 (0.00)
  Baseline - Bad Taste/change of taste | 0.0 (0.00) | 0.0 (0.00)
  Baseline - Headache | 0.1 (0.24) | 0.1 (0.23)
  Baseline - Fatigue Malaise | 0.2 (0.44) | 0.1 (0.32)
  Visit 2- Burning/Stinging Upon Instillation | 0.02 (0.39) | 0.2 (0.42)
  Visit 2- Non-Instillation Burning/Stinging | 0.0 (0.0) | 0.1 (0.32)
  Visit 2- Dry/Gritty Eye | 0.1 (0.33) | 0.2 (0.37)
  Visit 2- Foreign Body Sensation | 0.1 (0.49) | 0.1 (0.23)
  Visit 2- Eye Redness | 0.1 (0.24) | 0.1 (0.23)
  Visit 2- Blurred Vision | 0.0 (0.0) | 0.2 (0.37)
  Visit 2- Dry Mouth | 0.2 (0.53) | 0.3 (0.67)
  Visit 2- Bad Taste/Change of Taste | 0.0 (0.0) | 0.3 (0.65)
  Visit 2- Headache | 0.0 (0.0) | 0.0 (0.0)
  Visit 2- Fatique Malaise | 0.1 (0.33) | 0.0 (0.0)
  Visit 3- Burning/Stinging Upon Instillation | 0.4 (0.49) | 0.3 (0.58)
  Visit 3- Non-Instillation Burning/Stinging | 0.1 (0.24) | 0.1 (0.23)
  Visit 3- Dry/Gritty Eye | 0.2 (0.56) | 0.3 (0.67)
  Visit 3- Foreign Body Sensation | 0.1 (0.24) | 0.0 (0.0)
  Visit 3- Eye Redness | 0.1 (0.24) | 0.0 (0.0)
  Visit 3- Blurred Vision | 0.0 (0.0) | 0.0 (0.0)
  Visit 3- Dry Mouth | 0.2 (0.44) | 0.6 (0.96)
  Visit 3- Bad Taste/Change of Taste | 0.0 (0.0) | 0.4 (0.68)
  Visit 3- Headache | 0.1 (0.24) | 0.0 (0.0)
  Visit 3- Fatigue Malaise | 0.0 (0.0) | 0.1 (0.23)
  Visit 4- Burning/Stinging Upon Instillation | 0.4 (0.50) | 0.6 (0.80)
  Visit 4- Non-Instillation Burning/Stinging | 0.0 (0.0) | 0.1 (0.24)
  Visit 4- Dry/Gritty Eye | 0.2 (0.40) | 0.4 (0.61)
  Visit 4- Foreign Body Sensation | 0.0 (0.0) | 0.1 (0.33)
  Visit 4- Eye Redness | 0.2 (0.40) | 0.2 (0.73)
  Visit 4- Blurred Vision | 0.1 (0.25) | 0.1 (0.24)
  Visit 4- Dry Mouth | 0.4 (0.73) | 0.4 (0.71)
  Visit 4- Bad Taste/Change of Taste | 0.0 (0.0) | 0.3 (0.47)
  Visit 4- Headache | 0.0 (0.0) | 0.1 (0.33)
  Visit 4- Fatigue Malaise | 0.0 (0.0) | 0.1 (0.24)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time patients signed consent to their study exit, which was approximately 90 days for each patient.
Description: Site utilized a systematic assessment of adverse events on this trial. Adverse events (AEs) were assessed at each study visit outlined on the protocol. Subjects were instructed to contact site to report any AEs between study visits. Unscheduled visits were conducted to assess these reported AEs between study visits.
Arm/Group | Combigan BID | Simbrinza TID
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 3/21 | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combigan BID (N=21) | Simbrinza TID (N=22)
Ocular Adverse Events (Eye disorders) | 1 (1) | 2 (2)
Non-ocular Adverse Events (General disorders) | 2 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
The Local IRB closed in the middle of this trial which resulted in the discontinuation of 6 subjects. A new IRB was obtained and the study was re-opened and completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor may request but cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT02167035/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT02167035/SAP_001.pdf